CLINICAL TRIAL: NCT06860399
Title: The Effectiveness of Vardenafil Vs Sildenafil for The Treatment of Pulmonary Hypertension of the Newborn
Brief Title: Vardenafil Vs Sildenafil for the Treatment of Pulmonary Hypertension of the Newborn
Acronym: PPHN
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UDMS-Pediatrics-2025-01; 20230501 (Other: Damascus University)
Record Dates: First submitted 2025-02-19; First posted 2025-03-06 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: PPHN
Keywords: PPHN; Sildenafil; Vardenafil
MeSH Terms: interventions — Vardenafil Dihydrochloride; Sildenafil Citrate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vardenfil (Experimental): Oral Vardenafil given q12h.
  Interventions: Drug: Vardenafil
- Sildenafil (Active Comparator): Oral Sildenafil given q6h.
  Interventions: Drug: Sildenafil

INTERVENTIONS:
Drug: Vardenafil — Oral Vardenafil
  Other Names: fast fix
  Arms: Vardenfil
Drug: Sildenafil — Oral Sildenafil
  Other Names: viagra
  Arms: Sildenafil

SUMMARY:
The goal of this clinical trial is to learn if drug Vardenafil works to treat pulmonary hypertension in newborns, It will also learn about the safety of Vardenafil. The main questions it aims to answer are:

Does Vardenafil lower the pulmonary hypertension in newborns? What medical problems do participants have when taking Vardenafil? Researchers will compare drug Vardenafil to drug Sildenafil to see if drug Vardenafil works better to treat pulmonary hypertension.

Participants will be divided into 2 groups , one group will take oral drug: Vardenafil and the other group will take oral drug: Sildenafil every day.

Pulmonary hypertension will be measured daily until it returns to normal. Keep a diary of the symptoms and any complications

DETAILED DESCRIPTION:
A double blind controlled trial in Children's Hospital Damascus between 5/2023 and 9/2024 on newborns up to 4 d old diagnosed with PPHN, patients were allocated randomly into one of the 2 arms of the study, group Sildenafil and group Vardenafil, both medicines administered orally, management of the patients was the same in both groups except for the investigated drug, pulmonary hypertension and resistance were measured by echo at diagnosis time and every 24 hours later on till normalization of pulmonary pressure, at the end of recruitment data was collected and analyzed to confirm the safety of Vardenafil and compare the efficacy of Vardenafil to Sildenafil

ELIGIBILITY:
Inclusion Criteria:

* Gestation age: 28 weeks or more

Exclusion Criteria:

* Cardiac deformity, inability to administer the drug orally

Ages: 24 Hours to 96 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 55 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Pulmonary Hypertension | Pulmonary hypertension is evaluated for each participant at time of diagnosis before taking the drug = day 0, then every 24 hours until obtaining normal measurement (up to day 4)
  Pulmonary artery pressure is estimated from the tricuspid regurgitation velocity time measurement using echo doppler.
Pulmonary Resistance | Pulmonary resistance is evaluated for each participant at time of diagnosis before taking the drug = day 0, then every 24 hours until obtaining normal measurement (up to day 4)
  Echo measurement using pulmonary artery acceleration time to right ventricle ejection time ratio

SECONDARY OUTCOMES:
Respiratory Distress | Each participant is examined every 6 hours from time of diagnosis before taking the drug = day 0 until pulmonary pressure normalization (up to day 4)
  Respiratory rate and retractions evaluated by physical examination
Death | From day 1 of treatment till discharge from NICU ( 3 days to 90 days)

CONTACTS AND LOCATIONS:
Overall Officials: prof. Srour, Study Chair — Children's Hospital Damascus
Locations (1):
- Children's Hospital, Damascus, Syria

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, CSR
Time Frame: When summary data are published
Access Criteria: researchers working on the same topic interested in conducting the same study in different conditions or comparing the treatment to a different drug can contact the researcher by email